CLINICAL TRIAL: NCT03664063
Title: A Pharmacokinetic and Pharmacodynamic Evaluation of Co-Administration of IDA (Ivermectin, Diethylcarbamazine and Albendazole) & Azithromycin for Integrated Treatment of Neglected Tropical Diseases
Brief Title: PK PD Study of IDA and Azithromycin for NTDs ( ComboNTDs )
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lihir Medical Centre (Other)
Responsible Party: Principal Investigator, Oriol Mitja, Associate Professor, Lihir Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ComboNTDs-PK
Record Dates: First submitted 2018-09-03; First posted 2018-09-10 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Lymphatic Filariasis; Yaws; Trauma
MeSH Terms: conditions — Elephantiasis, Filarial; Yaws; Wounds and Injuries | interventions — Azithromycin; Albendazole; Ivermectin; Diethylcarbamazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Azithromycin for Yaws (Active Comparator): Patients will receive standard treatment for yaws alone
  Interventions: Drug: Azithromycin
- IDA for Lymphatic Filariasis (Active Comparator): Patients will receive standard IDA (Ivermectin & Diethylcarbamazine & Albendazole) treatment for Lymphatic Filariasis alone
  Interventions: Drug: Albendazole; Drug: Ivermectin; Drug: Diethylcarbamazine
- Combination Therapy of Azithromycin for Yaws and IDA for LF (Experimental): Patients will receive combination therapy for both yaws and IDA for Lymphatic Filariasis at the same time.
  Interventions: Drug: Azithromycin; Drug: Albendazole; Drug: Ivermectin; Drug: Diethylcarbamazine

INTERVENTIONS:
Drug: Azithromycin — Treatment with Azithromycin single dose - weight based dosing max 2gm
  Arms: Azithromycin for Yaws; Combination Therapy of Azithromycin for Yaws and IDA for LF
Drug: Albendazole — Single dose of Albendazole weight based dosing
  - 400mg
  Other Names: IDA
  Arms: Combination Therapy of Azithromycin for Yaws and IDA for LF; IDA for Lymphatic Filariasis
Drug: Ivermectin — Ivermectin weight based dosing - max 21mg
  Other Names: IDA
  Arms: Combination Therapy of Azithromycin for Yaws and IDA for LF; IDA for Lymphatic Filariasis
Drug: Diethylcarbamazine — Diethylcarbamazine weight based dosing - max 500mg
  Other Names: IDA
  Arms: Combination Therapy of Azithromycin for Yaws and IDA for LF; IDA for Lymphatic Filariasis

SUMMARY:
This is a Pharmacokinetic and Pharmacodynamic study evaluating the safety of co-administering Azithromycin alongside the new IDA (Ivermectin, Diethylcarbamazine, Albendazole) combination treatment for LF. Individuals will be randomised to receive Azithromycin alone, IDA or combination therapy. Clinical and biochemical monitoring for safety will be undertaken. Drug levels will be measured in each of the three arms to assess whether combination therapy significantly alters drug levels.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18-65
* Able to give informed consent

Exclusion Criteria:

* Known chronic illness
* Hb <7 at baseline
* Liver function or Creatinine * 1.5 Upper Limit of Normal
* Urinary tract infection at baseline
* Pregnancy (female participants only)
* Routine medications which interact with study drugs
* Lactose/Gluten intolerance
* Permanent disability impeding study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Drug levels of Azithromycin, Ivermectin, Diethylcarbamazine, Albendazole | 4 Days
  Plasma concentrations of Azithromycin, Ivermectin, Diethylcarbamize, Albendazole

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Four days
  Patients will undergo regular monitoring for the duration of the study - adverse events will be graded from 1 to 4 in line with the CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Lihir Medical Centre, Londolovit, New Ireland Province, Papua New Guinea

REFERENCES:
- [Derived] Alshehri A, Chhonker YS, Bala V, Edi C, Bjerum CM, Koudou BG, John LN, Mitja O, Marks M, King CL, Murry DJ. Population pharmacokinetic model of ivermectin in mass drug administration against lymphatic filariasis. PLoS Negl Trop Dis. 2023 Jun 1;17(6):e0011319. doi: 10.1371/journal.pntd.0011319. eCollection 2023 Jun. PMID 37262040
- [Derived] John LN, Bjerum C, Martinez PM, Likia R, Silus L, Wali C, Elizah A, Chhonker YS, Bala V, King CL, Murry DJ, Mitja O, Marks M. Pharmacokinetic and safety study of co-administration of albendazole, diethylcarbamazine, Ivermectin and azithromycin for the integrated treatment of Neglected Tropical Diseases. Clin Infect Dis. 2020 Aug 20:ciaa1202. doi: 10.1093/cid/ciaa1202. Online ahead of print. PMID 32818264